CLINICAL TRIAL: NCT02877264
Title: A Randomized, Single-Center, Open-Label, Three-Period, Six-Sequence, Crossover, Comparative Study to Compare the Oral Bioavailability of Single Doses of Three Vapendavir Drug Product Formulations in Healthy Volunteers
Brief Title: A Study to Compare the Oral Bioavailability of Single Doses of Three Vapendavir Drug Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aviragen Therapeutics (Industry)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BTA798-104
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Vapendavir; Bioavailability; Biological Availability; Volunteers
MeSH Terms: interventions — Tablets; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vapendavir Capsule, 264 mg (Experimental): Vapendavir phosphate salt administered orally as a single dose of two 132 mg hard gelatin capsules
  Interventions: Drug: vapendavir 132 mg capsule
- Vapendavir Tablets, 264 mg (Experimental): Vapendavir free base tablets containing 264 mg of vapendavir
  Interventions: Drug: vapendavir 264 mg tablet
- Vapendavir Oral Suspension, 264 mg (Experimental): Vapendavir free base as a 24 mg/mL oral suspension
  Interventions: Drug: vapendavir 24 mg/mL oral suspension

INTERVENTIONS:
Drug: vapendavir 132 mg capsule
  Other Names: BTA798
  Arms: Vapendavir Capsule, 264 mg
Drug: vapendavir 264 mg tablet
  Other Names: BTA798
  Arms: Vapendavir Tablets, 264 mg
Drug: vapendavir 24 mg/mL oral suspension
  Other Names: BTA798
  Arms: Vapendavir Oral Suspension, 264 mg

SUMMARY:
This is a randomized, single-center, open-label, three-period, six-sequence, crossover, comparative study to evaluate the oral bioavailability of single doses of three vapendavir drug product formulations (the 264 mg free base tablet [test drug], 264 mg free base oral suspension [test drug], and two 132 mg phosphate salt capsules [reference drug]) in healthy volunteers. The study design consists of six dosing sequences. Each sequence comprises 3 periods and each subject is administered one of the three dosing formulations in the first period. A subject receives a different formulation in each of the subsequent periods, so that all subjects receive each formulation. The periods are separated by an approximate 7-day washout.

DETAILED DESCRIPTION:
Owner of Study Record: Vaxart Inc.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a healthy male or female between 19 and 60 years of age (inclusive) at the time of signing the informed consent and weigh ≥50 kg with a BMI between 18 and 32.0 kg/m2 (inclusive);
2. Capable of giving written informed consent;
3. Subject is able to understand and comply with the protocol requirements, instructions and restrictions;
4. Healthy on the basis of physical examination, medical history, VS, ECGs, and clinical laboratory tests;
5. Female subjects who are not postmenopausal for at least 2 years or surgically sterile with complete hysterectomy or bilateral oophorectomy and male subjects, who are not surgically sterile via vasectomy, must agree to use a double barrier method of birth control, such as, a condom plus spermicidal agent (foam/gel/film/cream/suppository) from Study Day 0 until 30 days after completion of the study. This includes female subjects who are using hormonal contraception;
6. Female subjects must not be breastfeeding or pregnant.

Exclusion Criteria:

1. Positive results at screening for hepatitis B, hepatitis C, or HIV;
2. No use of tobacco products, as well as electronic cigarettes, within 14 days of Study Day 1 or unwilling to abstain during study participation;
3. A medical history or clinical evidence of any clinical condition that may, in the opinion of the Investigator or Medical Monitor, impact on the subject's ability to participate in the study, or on the study results;
4. Current or recent respiratory or other infection within 14 days of screening;
5. Presence or history of significant allergy requiring treatment;
6. Clinically significant abnormalities on ECG;
7. Vital signs representing abnormal systolic blood pressure and/or abnormal diastolic blood pressure;
8. Safety laboratory abnormalities at screening or Study Day 0 which are clinically significant;
9. Subject has a history of drug abuse or alcohol abuse in the past 2 years or current evidence of such abuse or addiction;
10. A positive urine drug screen test at screening or admission to the study facility;
11. A positive breathalyzer for alcohol at screening or admission to the study facility;
12. A positive pregnancy test at screening or admission to the study facility;
13. Abstinence from alcohol must be employed from 72 hours before Study Day 1 and throughout the duration of study participation;
14. Use of chronic prescription medications within 90 days, with the exception of hormonal contraceptives (or contraceptive device containing hormonal contraceptive) being taken by female subjects within 14 days, or over-the-counter (OTC) medications, including vitamin, herbal, and mineral supplements, within the 7 days prior to Study Day 1 and throughout study participation;
15. Received an investigational drug or investigational vaccine within 30 days, or use of an investigational medical device within 30 days prior to Study Day 1;
16. Any prior use of vapendavir or inclusion in a previous vapendavir investigational study or ongoing participation in a vapendavir investigational study;
17. Donation or loss of whole blood within 60 days or plasma within 14 days of Study Day 1 or anytime from screening to 30 days after completion of the study.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Relative oral bioavailability, as applicable | Study Day 0 - 17
Maximum observed plasma concentration (Cmax) | Study Day 0 - 17
Time at which Cmac was observed (Tmax) | Study Day 0 - 17
Area under the plasma concentration time curve from time ) to the last measureable plasma concentration (AUC 0-last) | Study Day 0 - 17

CONTACTS AND LOCATIONS:
Overall Officials: Anna Novotney-Barry, Study Director — Aviragen Therapeutics, Inc.
Locations (1):
- Aviragen Investigational Site, Saint Paul, Minnesota, United States